CLINICAL TRIAL: NCT01628549
Title: A Randomized, Multicenter, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of 3 Different Doses of a Novel Tetracycline Compared to Placebo in the Treatment of Facial Acne Vulgaris, Study PR-10411
Brief Title: Double-Blind, Placebo-Controlled Study to Evaluate 3 Doses of a Novel Tetracycline in the Treatment of Facial Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PR-10411
Record Dates: First submitted 2012-06-22; First posted 2012-06-26 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Acne Vulgaris
Keywords: acne
MeSH Terms: conditions — Acne Vulgaris | interventions — sarecycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- P005672-HCl approximately 0.75 mg/kg/day (Experimental): One P005672-HCl 50 mg capsule and one Placebo capsule, oral administration, once daily for 12 weeks
  Interventions: Drug: 50 mg P005672-HCl; Drug: Placebo
- P005672-HCl approximately 1.5 mg/kg/day (Experimental): Two P005672-HCl 50mg capsules, oral administration, once daily for 12 weeks
  Interventions: Drug: 50 mg P005672-HCl
- P005672-HCl approximately 3.0 mg/kg/day (Experimental): Two P005672-HCl 100mg capsules, oral administration, once daily for 12 weeks
  Interventions: Drug: 100 mg P005672-HCl
- Placebo (Placebo Comparator): Two Placebo capsules matching P005672-HCl, oral administration, once daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 50 mg P005672-HCl — P005672-HCl administered as an oral capsule(s) once daily
  Other Names: WC3035, Sarecycline
  Arms: P005672-HCl approximately 0.75 mg/kg/day; P005672-HCl approximately 1.5 mg/kg/day
Drug: Placebo — Dose-matched Placebo capsule administered as an oral capsule(s) once daily
  Other Names: Inactive
  Arms: P005672-HCl approximately 0.75 mg/kg/day; Placebo
Drug: 100 mg P005672-HCl — P005672-HCl administered as an oral capsule(s) once daily
  Other Names: WC3035, Sarecycline
  Arms: P005672-HCl approximately 3.0 mg/kg/day

SUMMARY:
To evaluate the safety and effectiveness of 3 strengths of P005672-HCl compared to placebo for the treatment of moderate to severe facial acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* if women of child-bearing potential, have a negative urine pregnancy test
* Willing to use only a non-medicated cleanser and to refrain from use of any other acne medication, medicated cleanser, excessive sun exposure, and tanning booths for the duration of the study
* Male or female, 12-45 years of age with body weight between 52 and 88 kg
* Diagnosis of acne vulgaris with:

  20 to 50 inflammatory lesions (papules, pustules, and nodules) 30 to 100 noninflammatory lesions (open and closed comedones)
* No more than 2 nodules on the face
* Investigator's Global Assessment (IGA) score of moderate (3) to severe (4)

Exclusion Criteria:

* Dermatological condition of face or facial hair that could interfere with clinical evaluations subjects who have used the following medications (topical refers only to the facial area) will not be eligible:

Within 1 week prior to randomization:

* Medicated facial cleansers
* Topical acne treatments (other than those listed below)

Within 4 weeks prior to randomization:

* Topical retinoids
* Topical anti-inflammatories and corticosteroids
* Systemic antibiotics
* Systemic acne treatments

Within 12 weeks prior to randomization:

* Systemic retinoids
* Systemic corticosteroids
* Pseudomembranous colitis or antibiotic-associated colitis
* Hepatitis, liver damage or renal impairment

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 285 (Actual)
Dates: Start 2012-06-30 (Actual); Primary Completion 2012-11-16 (Actual); Study Completion 2013-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herman Ellman, MD, Study Director — Warner Chilcott
Locations (37):
- United States (37):
  - Warner Chilcott Investigational Site, Mobile, Alabama
  - Warner Chilcott Investigational Site, Tucson, Arizona
  - Warner Chilcott Investigational Site, Hot Springs, Arkansas
  - Warner Chilcott Investigational Site, Los Angeles, California
  - Warner Chilcott Investigational Site, San Diego, California
  - Warner Chilcott Investigational Site, Santa Monica, California
  - Warner Chilcott Investigational Site, Clearwater, Florida
  - Warner Chilcott Investigational Site, Coral Gables, Florida
  - Warner Chilcott Investigational Site, Gainesville, Florida
  - Warner Chilcott Investigational Site, Miami, Florida
  - Warner Chilcott Investigational Site, Miramar, Florida
  - Warner Chilcott Investigational Site, Pinellas Park, Florida
  - Warner Chilcott Investigational Site, Arlington Heights, Illinois
  - Warner Chilcott Investigational Site, Chicago, Illinois
  - Warner Chilcott Investigational Site, Granger, Indiana
  - Warner Chilcott Investigational Site, Indianapolis, Indiana
  - Warner Chilcott Investigational Site, Louisville, Kentucky
  - Warner Chilcott Investigational Site, Boston, Massachusetts
  - Warner Chilcott Investigational Site, Fridley, Minnesota
  - Warner Chilcott Investigational Site, St Louis, Missouri
  - Warner Chilcott Investigational Site, Berlin, New Jersey
  - Warner Chilcott Investigational Site, Albuquerque, New Mexico
  - Warner Chilcott Investigational Site, Rochester, New York
  - Warner Chilcott Investigational Site, Charlotte, North Carolina
  - Warner Chilcott Investigational Site, Salisbury, North Carolina
  - Warner Chilcott Investigational Site, Wilmington, North Carolina
  - Warner Chilcott Investigational Site, Cincinnati, Ohio
  - Warner Chilcott Investigational Site, Portland, Oregon
  - Warner Chilcott Investigational Site, Philadelphia, Pennsylvania
  - Warner Chilcott Investigational Site, Greer, South Carolina
  - Warner Chilcott Investigational Site, Arlington, Texas
  - Warner Chilcott Investigational Site, Austin, Texas
  - Warner Chilcott Investigational Site, Houston, Texas
  - Warner Chilcott Investigational Site, Plano, Texas
  - Warner Chilcott Investigational Site, San Antonio, Texas
  - Warner Chilcott Investigational Site, Sandy City, Utah
  - Warner Chilcott Investigational Site, Lynchburg, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Two placebo capsules matching P005672-HCl, taken orally each day
- P005672-HCl Approximately 0.75 mg/kg/Day: One P005672-HCl 50 mg capsule and one Placebo capsule, taken orally each day
- P005672-HCl Approximately 1.5 mg/kg/Day: Two P005672-HCl 50 mg capsules, taken orally each day
- P005672-HCl Approximately 3.0 mg/kg/Day: Two P005672-HCl 100 mg capsules, taken orally each day
Period: Overall Study
Arm/Group | Placebo | P005672-HCl Approximately 0.75 mg/kg/Day | P005672-HCl Approximately 1.5 mg/kg/Day | P005672-HCl Approximately 3.0 mg/kg/Day
Started | 73 | 76 | 70 | 66
Completed | 64 | 64 | 60 | 57
Not Completed | 9 | 12 | 10 | 9
Not completed — Adverse Event | 1 | 1 | 0 | 4
Not completed — Lost to Follow-up | 3 | 4 | 3 | 3
Not completed — Withdrawal by Subject | 3 | 4 | 4 | 1
Not completed — Protocol Violation | 2 | 1 | 1 | 0
Not completed — withdrawn for noncompliance | 0 | 2 | 1 | 0
Not completed — abnormal laboratory test results | 0 | 0 | 1 | 0
Not completed — positive pregnancy test | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: 285 participants were randomized to double-blind treatment (Safety population)
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | P005672-HCl Approximately 0.75 mg/kg/Day | P005672-HCl Approximately 1.5 mg/kg/Day | P005672-HCl Approximately 3.0 mg/kg/Day | Total
Number analyzed (Participants) | 73 | 76 | 70 | 66 | 285
Age, Continuous [Mean (Standard Deviation); unit: Years] | 20.8 (6.99) | 19.7 (5.92) | 19.9 (7.04) | 20.3 (7.11) | 20.2 (6.74)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 25 | 29 | 30 | 29 | 113
  Female | 48 | 47 | 40 | 37 | 172
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 19 | 21 | 16 | 19 | 75
  Not Hispanic or Latino | 54 | 55 | 54 | 47 | 210
Race/Ethnicity, Customized [Number; unit: Participants] — Population: Five subjects in the Safety Population checked multiple races.
  Participants
    American Indian or Alaska Native | 1 | 0 | 0 | 1 | 2
    Asian | 4 | 4 | 3 | 1 | 12
    Black or African American | 17 | 18 | 21 | 13 | 69
    Native Hawaiian or Other Pacific islander | 0 | 0 | 0 | 0 | 0
    White | 54 | 55 | 46 | 52 | 207
Height [Mean (Standard Deviation); unit: cm] | 165.80 (10.436) | 167.49 (9.047) | 167.23 (7.380) | 167.33 (9.764) | 166.96 (9.206)
Weight at Baseline [Mean (Standard Deviation); unit: kg] | 68.47 (10.306) | 66.37 (8.749) | 69.69 (11.861) | 67.31 (9.486) | 67.94 (10.173)

OUTCOME MEASURES:

1. Primary Outcome: The Absolute Change From Baseline in the Inflammatory Lesion Count at the Final Visit
Time Frame: Baseline (Week 0) to Final Visit (Up to Week 12)
Population: Of the 285 participants in the Safety Population, 284 received a post-Baseline efficacy assessment, to comprise the mITT (Modified Intent-to-Treat) Population.
Measure: Mean (Standard Deviation); unit: Number of Inflammatory Lesions
Arm/Group | Placebo | P005672-HCl Approximately 0.75 mg/kg/Day | P005672-HCl Approximately 1.5 mg/kg/Day | P005672-HCl Approximately 3.0 mg/kg/Day
Number analyzed (Participants) | 72 | 76 | 70 | 66
Number of Inflammatory Lesions | 12.8 (14.18) | 14.4 (13.01) | 17.6 (16.65) | 17.1 (11.69)
Statistical Analysis 1: Comparison: Placebo vs P005672-HCl Approximately 0.75 mg/kg/Day; Test type: Superiority; p = 0.4344, ANCOVA; Difference in Least Squares Means = 1.53, 95% CI 2-sided [-2.32 to 5.38]
Statistical Analysis 2: Comparison: Placebo vs P005672-HCl Approximately 1.5 mg/kg/Day; Test type: Superiority; p = 0.0266, ANCOVA; Difference in Least Squares Means = 4.46, 95% CI 2-sided [0.52 to 8.40]
Statistical Analysis 3: Comparison: Placebo vs P005672-HCl Approximately 3.0 mg/kg/Day; Test type: Superiority; p = 0.0317, ANCOVA; Difference in Least Squares Means = 4.37, 95% CI 2-sided [0.39 to 8.36]

2. Primary Outcome: The Dichotomized IGA (Investigator Global Assessment) Score at Final Visit
Description: The Investigator Global Assessment Scale (IGA) for Acne Vulgaris Score is a 5-point ordinal scale ranging from 0 to 4.
  The dichotomized IGA score, where success was defined as at least a 2-grade decrease in the IGA score during the Final Visit as compared to the Baseline Visit.
Time Frame: Final Visit (Up to Week 12)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | P005672-HCl Approximately 0.75 mg/kg/Day | P005672-HCl Approximately 1.5 mg/kg/Day | P005672-HCl Approximately 3.0 mg/kg/Day
Number analyzed (Participants) | 72 | 76 | 70 | 66
Participants
  Success | 8 | 11 | 17 | 10
  Failure | 64 | 65 | 53 | 56
Statistical Analysis 1: Comparison: Placebo vs P005672-HCl Approximately 0.75 mg/kg/Day; Test type: Superiority; p = 0.3300, Cochran-Mantel-Haenszel; Difference vs placebo in success rate = 3.4, 95% CI 2-sided [-7.82 to 14.38]
Statistical Analysis 2: Comparison: Placebo vs P005672-HCl Approximately 1.5 mg/kg/Day; Test type: Superiority; p = 0.0159, Cochran-Mantel-Haenszel; Difference vs placebo in success rate = 13.2, 95% CI 2-sided [0.54 to 25.60]
Statistical Analysis 3: Comparison: Placebo vs P005672-HCl Approximately 3.0 mg/kg/Day; Test type: Superiority; p = 0.4834, Cochran-Mantel-Haenszel; Difference vs placebo in success rate = 4.1, 95% CI 2-sided [-7.44 to 15.87]

3. Secondary Outcome: The Absolute Change From Baseline in the Inflammatory Lesion Count at Weeks 1, 2, 4, 8, 12 and the Final Visit
Time Frame: Baseline (Week 0) up to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Count of Inflammatory Lesions
Arm/Group | Placebo | P005672-HCl Approximately 0.75 mg/kg/Day | P005672-HCl Approximately 1.5 mg/kg/Day | P005672-HCl Approximately 3.0 mg/kg/Day
Number analyzed (Participants) | 72 | 76 | 70 | 66
Count of Inflammatory Lesions
  Change from Baseline at Week 1 | 5.8 (9.07) | 5.4 (9.28) | 5.4 (8.44) | 5.9 (8.33)
  Change from Baseline at Week 2 | 8.4 (10.13) | 8.5 (10.02) | 8.2 (14.45) | 9.7 (11.30)
  Change from Baseline at Week 4 | 10.9 (10.04) | 9.3 (13.84) | 11.7 (15.36) | 12.8 (9.96)
  Change from Baseline at Week 8 | 12.6 (12.57) | 13.1 (11.89) | 15.0 (16.66) | 14.3 (12.90)
  Change from Baseline at Week 12 | 12.8 (14.18) | 14.3 (13.00) | 17.6 (16.65) | 17.1 (11.69)
  Change from Baseline at Final Visit(Up to Week 12) | 12.8 (14.18) | 14.4 (13.01) | 17.6 (16.65) | 17.1 (11.69)

4. Secondary Outcome: The Absolute Change From Baseline in the Noninflammatory Lesion Count at Weeks 1, 2, 4, 8, 12, and the Final Visit
Time Frame: Baseline (Week 0) up to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Count of Noninflammatory Lesions
Arm/Group | Placebo | P005672-HCl Approximately 0.75 mg/kg/Day | P005672-HCl Approximately 1.5 mg/kg/Day | P005672-HCl Approximately 3.0 mg/kg/Day
Number analyzed (Participants) | 72 | 76 | 70 | 66
Count of Noninflammatory Lesions
  Change from Baseline at Week 1 | 5.4 (12.99) | 3.8 (14.28) | 4.3 (14.10) | 5.1 (13.83)
  Change from Baseline at Week 2 | 10.6 (16.02) | 9.4 (13.58) | 7.8 (16.92) | 7.9 (14.24)
  Change from Baseline at Week 4 | 13.0 (24.17) | 10.0 (17.25) | 9.9 (20.58) | 12.7 (15.24)
  Change from Baseline at Week 8 | 16.9 (22.52) | 14.3 (21.44) | 14.0 (22.22) | 15.2 (19.04)
  Change from Baseline at Week 12 | 17.8 (21.63) | 17.9 (19.85) | 19.1 (22.33) | 17.0 (21.56)
  Change from Baseline at Final Visit(Up to Week 12) | 17.8 (21.63) | 17.9 (19.83) | 19.1 (22.33) | 17.0 (21.56)

5. Secondary Outcome: The Percent Change From Baseline in the Inflammatory Lesion Count at Weeks 1, 2, 4, 8, 12, and the Final Visit
Time Frame: Baseline (Week 0) up to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change - Inflammatory Lesions
Arm/Group | Placebo | P005672-HCl Approximately 0.75 mg/kg/Day | P005672-HCl Approximately 1.5 mg/kg/Day | P005672-HCl Approximately 3.0 mg/kg/Day
Number analyzed (Participants) | 72 | 76 | 70 | 66
Percent Change - Inflammatory Lesions
  Change from Baseline at Week 1 | 19.3 (27.82) | 17.2 (28.43) | 17.8 (26.39) | 19.4 (26.17)
  Change from Baseline at Week 2 | 25.6 (29.02) | 26.4 (32.60) | 25.8 (36.16) | 30.6 (35.88)
  Change from Baseline at Week 4 | 34.1 (28.84) | 29.3 (38.90) | 34.1 (35.27) | 40.0 (31.83)
  Change from Baseline at Week 8 | 37.9 (35.60) | 39.8 (34.47) | 44.3 (37.99) | 44.5 (37.62)
  Change from Baseline at Week 12 | 39.1 (43.00) | 43.3 (39.70) | 53.6 (37.65) | 53.5 (35.18)
  Change from Baseline at Final Visit(Up to Week 12) | 39.1 (43.00) | 43.5 (39.72) | 53.6 (37.65) | 53.5 (35.18)

6. Secondary Outcome: The Percent Change From Baseline in the Noninflammatory Lesion Count at Weeks 1, 2, 4, 8, 12, and the Final Visit
Time Frame: Baseline (Week 0) up to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change - noninflammatory lesions
Arm/Group | Placebo | P005672-HCl Approximately 0.75 mg/kg/Day | P005672-HCl Approximately 1.5 mg/kg/Day | P005672-HCl Approximately 3.0 mg/kg/Day
Number analyzed (Participants) | 72 | 76 | 70 | 66
Percent change - noninflammatory lesions
  Change from Baseline at Week 1 | 9.7 (24.07) | 7.7 (26.87) | 8.3 (25.20) | 10.6 (25.63)
  Change from Baseline at Week 2 | 19.0 (28.36) | 16.7 (24.99) | 14.6 (30.57) | 16.0 (30.37)
  Change from Baseline at Week 4 | 25.0 (37.78) | 18.3 (33.17) | 19.2 (35.60) | 25.7 (29.27)
  Change from Baseline at Week 8 | 30.5 (40.69) | 26.1 (38.84) | 27.5 (38.54) | 30.4 (38.45)
  Change from Baseline at Week 12 | 35.3 (35.32) | 34.3 (36.40) | 37.2 (38.44) | 32.8 (42.59)
  Change from Baseline at Final Visit(Up to Week 12) | 35.3 (35.32) | 34.1 (36.28) | 37.2 (38.44) | 32.8 (42.59)

7. Secondary Outcome: The Dichotomized IGA Score at Weeks 1, 2, 4, 8, and 12
Description: as for outcome 2
Time Frame: Baseline to Final Visit (Up to Week 12)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | P005672-HCl Approximately 0.75 mg/kg/Day | P005672-HCl Approximately 1.5 mg/kg/Day | P005672-HCl Approximately 3.0 mg/kg/Day
Number analyzed (Participants) | 72 | 76 | 70 | 66
Participants
  Week 1: Success | 0 | 3 | 0 | 1
  Week 1: Failure | 72 | 73 | 70 | 65
  Week 2: Success | 2 | 3 | 2 | 2
  Week 2: Failure | 70 | 73 | 68 | 64
  Week 4: Success | 1 | 2 | 0 | 4
  Week 4: Failure | 71 | 74 | 70 | 62
  Week 8: Success | 6 | 6 | 8 | 11
  Week 8: Failure | 66 | 70 | 62 | 55
  Week 12: Success | 8 | 11 | 17 | 10
  Week 12: Failure | 64 | 65 | 53 | 56
  Final Visit (Up to Week 12): Success | 8 | 11 | 17 | 10
  Final Visit (Up to Week 12): Failure | 64 | 65 | 53 | 56

ADVERSE EVENTS:
Time Frame: From Screening (up to week -12) to Week 12 plus 30 days.
Arm/Group | Placebo | P005672-HCl Approximately 0.75 mg/kg/Day | P005672-HCl Approximately 1.5 mg/kg/Day | P005672-HCl Approximately 3.0 mg/kg/Day
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/76 | 0/70 | 0/66
Other Adverse Events (participants affected / at risk) | 13/73 | 15/76 | 8/70 | 7/66
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=73) | P005672-HCl Approximately 0.75 mg/kg/Day (N=76) | P005672-HCl Approximately 1.5 mg/kg/Day (N=70) | P005672-HCl Approximately 3.0 mg/kg/Day (N=66)
Headache (Nervous system disorders) | 8 | 5 | 5 | 4
Nausea (Gastrointestinal disorders) | 4 | 6 | 1 | 2
Nasopharyngitis (Infections and infestations) | 5 | 4 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The data obtained in this study are the property of the Sponsor, any manuscript or other presentation of data must first be reviewed by the Sponsor before its submission.